CLINICAL TRIAL: NCT03331393
Title: The Value of Orencia in Rapidly Progressing Rheumatoid Arthritis: A Chart Review Study
Brief Title: The Value of Orencia in Rapidly Progressing Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-686
Record Dates: First submitted 2017-10-17; First posted 2017-11-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RA patients treated with Abatacept: Treated with Abatacept as a first-line biologic
  Interventions: Other: Non-interventional
- RA patients treated with TNFi: Treated with Tumor necrosis factor inhibitor (TNFi) as a first-line biologic
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — Non-interventional

SUMMARY:
The purpose of this study is to investigate the value of Orencia in rapidly progressing Rheumatoid Arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age at enrollment
* Confirmed diagnosed with RA
* Initiated first-line treatment with abatacept, adalimumab, etanercept, or infliximab with a record of the start date at the practice site

Exclusion Criteria:

* Does not have at least 1 or more poor RA prognostic factor: Evidence of joint erosions, Positive anti-CCP autoantibodies, Positive RF autoantibodies, Increased CRP levels, Increased ESR levels
* Was followed at the site for less than 1 year since biologic treatment initiation
* Patients with autoimmune diseases: Crohn's, ankylosing spondylitis, ulcerative colitis, psoriatic arthritis, anal fistula

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rapidly-progressing RA patients initiating treatment with abatacept or TNFi at approximately 10 rheumatology practices across the US.
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
number of patients discontinuing treatment before completing 12 months of therapy | approximately 1 year
time from treatment initiation to discontinuation | approximately 1 year

SECONDARY OUTCOMES:
Distribution of Healthcare Resource Utilization (HCRU) | approximately 1 year
Disease Activity Score | approximately 1 year
  Disease Activity Score (DAS)
Health Assessment Questionnaire | approximately 1 year
  Health Assessment Questionnaire (HAQ)
C-reactive Protein Levels | approximately 1 year
  C-reactive protein (CRP) levels
Erythrocyte Sedimentation Rate | approximately 1 year
  Erythrocyte sedimentation rate (ESR) levels
Joint Erosions | approximately 1 year
  Measured by radiographic reports

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- United States (7):
  - Local Institution, Beverly Hills, California
  - Local Institution - 0005, Gainesville, Georgia
  - Local Institution, Coeur d'Alene, Idaho
  - Local Institution - 0007, Eagan, Minnesota
  - Medication Management, LLC, Greensboro, North Carolina
  - Local Institution, Myrtle Beach, South Carolina
  - Local Institution, Richland, Washington

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm